CLINICAL TRIAL: NCT01192633
Title: Phase Ⅱ Study of Gemcitabine,Vincristine and Cisplatin as Second Line Combination Therapy in Patients With Sarcoma
Brief Title: Gemcitabine,Vincristine and Cisplatin as Second Line Combination Therapy in Patients With Sarcoma
Acronym: GVPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GVP-SAR
Record Dates: First submitted 2010-03-25; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Sarcoma; Chemotherapy
Keywords: Sarcoma; gemcitabine; vincristine; cisplatin; chemotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GVP — Drug: gemcitabine, vincristine,cisplatin
  cisplatin 25mg/m2，ivgtt，D1, 2, 3 gemcitabine 1000mg/m2，ivgtt，30'，D1, 8 vincristine 1.4mg/m2(less than 2 mg), iv, D1 repeat every 3 weeks

SUMMARY:
The primary objective of this study is to evaluate PFS of gemcitabine,vincristine and cisplatin as second line therapy in patients with sarcoma. 40 patients will be treated into this study.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent prior to study, with understanding that the patient has the right to withdraw from the study at any time without prejudice
* Be female of male and ≥18 and ≤75 years of age
* Be ambulatory and have ECOG performance status of ≤1
* Have histological confirmed sarcoma
* Locally advanced or metastatic sarcoma who receive first-line chemotherapy.
* Have at least one target lesion according to the RECIST criteria.

Exclusion Criteria:

* Pregnant or lactating women
* patient has received chemotherapy drugs including gemcitabine,vincristine and cisplatin
* Chemotherapy within four weeks preceding treatment start
* ECOG ≥ 2
* Radiotherapy to the axial skeleton within the 4 weeks preceding study treatment start or insufficient recovery from the effects of prior radiotherapy
* Participation in any investigational drug study within 4 weeks preceding treatment start
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix .Abnormal laboratory values: hemoglobin < 8. 0g/dl, neutrophil< 1.5×109/L, platelet< 100×109/L.
* serum creatine > upper limit of normal (ULN)
* serum bilirubin > ULN
* alanine aminotransferase(ALT) and aspartate aminotransferase(AST)>5×ULN
* alkaline phosphatase(AKP)>5×ULN
* Serious uncontrolled intercurrence infection
* Life expectancy of less than 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(Progression-free survival was evaluated for the period from the date of first treatment with this regimen to the date when disease progression was first observed or death occurred.) | every 6 weeks

SECONDARY OUTCOMES:
Response Rate | every 6 weeks
Overall Survival | 2 years
Side Effects | every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Hong, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Patel SR, Gandhi V, Jenkins J, Papadopolous N, Burgess MA, Plager C, Plunkett W, Benjamin RS. Phase II clinical investigation of gemcitabine in advanced soft tissue sarcomas and window evaluation of dose rate on gemcitabine triphosphate accumulation. J Clin Oncol. 2001 Aug 1;19(15):3483-9. doi: 10.1200/JCO.2001.19.15.3483. PMID 11481354
- [Result] Hartmann JT, Oechsle K, Huober J, Jakob A, Azemar M, Horger M, Kanz L, Bokemeyer C. An open label, non-comparative phase II study of gemcitabine as salvage treatment for patients with pretreated adult type soft tissue sarcoma. Invest New Drugs. 2006 May;24(3):249-53. doi: 10.1007/s10637-005-3537-1. PMID 16133789
- [Derived] Luo Z, Zhang X, Peng W, Wu X, Wang H, Yu H, Wang J, Chang J, Hong X. A Phase II Study of Gemcitabine, Vincristine, and Cisplatin As Second-Line Treatment for Patients with Advanced Soft Tissue Sarcoma. Medicine (Baltimore). 2015 Oct;94(43):e1777. doi: 10.1097/MD.0000000000001777. PMID 26512574